CLINICAL TRIAL: NCT01215851
Title: A Phase II Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of the Following: TMC207 Alone, TMC207 Plus Pyrazinamide,TMC207 Plus PA-824,PA-824 Plus Pyrazinamide and PA-824 Plus Pyrazinamide and Moxifloxacin, in Adult Patients With Newly Diagnosed, Smear-Positive Pulmonary Tuberculosis.
Brief Title: Evaluation of Early Bactericidal Activity in Pulmonary Tuberculosis With(J-M-Pa-Z) (NC-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC-001-(J-M-Pa-Z)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; EBA; TMC207; pretomanid; Early Bactericidal Activity; Pulmonary Tuberculosis; PA-824; bedaquiline; pyrazinamide; moxifloxacin; ethambutol; rifafour
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — pretomanid; Pyrazinamide; bedaquiline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TMC207 (Experimental): TMC207 administered once daily as 100mg tablet for total daily dose of 700 mg on Day 1; 500mg on Day 2; 400mg on Days 3-14 plus pyrazinamide placebo administered once daily
  Interventions: Drug: TMC207
- TMC207 and pyrazinamide (Experimental): TMC207 administered once daily as 100mg tablet for total daily dose of 700 mg on Day 1; 500mg on Day 2; 400mg on Days 3-14 plus pyrazinamide administered once daily in 500mg tablets dosed by weight as follows: < or = 55kg received 2 tablets/day; >55kg to 75kg received 3 tablets/day; >75kg received 4 tablets/day
  Interventions: Drug: Pyrazinamide; Drug: TMC207
- PA-824 and pyrazinamide (Experimental): PA-824 administered once daily as 200mg tablets and pyrazinamide administered once daily in 500mg tablets dosed by weight as follows: < or = 55kg received 2 tablets/day; >55kg to 75kg received 3 tablets/day; >75kg received 4 tablets/day and moxifloxacin placebo (matched to moxifloxacin tablets) administered once daily
  Interventions: Drug: PA-824; Drug: Pyrazinamide
- PA-824 and moxifloxacin and pyrazinamide (Experimental): PA-824 administered once daily as 200mg tablets and pyrazinamide administered once daily in 500mg tablets dosed by weight as follows: < or = 55kg received 2 tablets/day; >55kg to 75kg received 3 tablets/day; >75kg received 4 tablets/day and moxifloxacin administered once daily as 400mg tablets
  Interventions: Drug: PA-824; Drug: Moxifloxacin
- Rifafour e-275 mg (Active Comparator): Rifafour e-275 administered once daily with each tablet containing 150mg rifampicin, 75mg isoniazid, 400mg pyrazinamide, and 275mg ethambutol and dose by weight as follows: 30kg-37kg received 2 tablets/day; 38kg-54kg received 3 tablets/days; 55kg-70kg received 4 tablets/day; > or = 71kg received 5 tablets/day
  Interventions: Drug: Rifafour
- TMC207 and PA-824 (Experimental): TMC207 administered once daily as 100mg tablet for total daily dose of 700 mg on Day 1; 500mg on Day 2; 400mg on Days 3-14 plus PA-824 administered once daily as 200mg tablets
  Interventions: Drug: PA-824; Drug: TMC207

INTERVENTIONS:
Drug: PA-824 — 200 mg tablet, once daily for 14 days
  Arms: PA-824 and moxifloxacin and pyrazinamide; PA-824 and pyrazinamide; TMC207 and PA-824
Drug: Pyrazinamide — Dosed by Weight
  Arms: PA-824 and pyrazinamide; TMC207 and pyrazinamide
Drug: TMC207 — TMC207 700 mg Day 1; 500mg Day 2; 400mg Days 3-14
  Arms: TMC207; TMC207 and PA-824; TMC207 and pyrazinamide
Drug: Rifafour — Rifafour e-275
  Arms: Rifafour e-275 mg
Drug: Moxifloxacin — moxifloxacin 400 mg
  Arms: PA-824 and moxifloxacin and pyrazinamide

SUMMARY:
The trial will evaluate the extended bactericidal activity of 14 consecutive days of oral administration of TMC207 alone, TMC207 with pyrazinamide, TMC207 with PA-824, PA-824 with pyrazinamide and PA-824 with moxifloxacin and pyrazinamide, as determined by the rate of change of log CFU in sputum over the time period Day 0-14 in participants with smear positive pulmonary tuberculosis (TB). A control group will receive standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, sputum smear-positive pulmonary TB.
5. A chest X-ray picture which in the opinion of the Investigator is compatible with TB.
6. Sputum positive on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale).
7. Ability to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).
8. Females may participate if they are: 1) of non-childbearing potential (have had a bilateral oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months), 2) if they are using effective birth control methods and are willing to continue practicing birth control methods throughout treatment or 3) be non-heterosexually active, practice sexual abstinence or have a vasectomized partner (confirmed sterile). Therefore to be eligible for this study women of childbearing potential should either: 1) use a double barrier method to prevent pregnancy (i.e. use a condom with either diaphragm or cervical cap) or 2) use hormonal based contraceptives in combination with a barrier contraceptive, or 3) use an intrauterine device in combination with a barrier contraceptive. They must also be willing to continue these contraceptive measures until 6 months after the last dose of study medication or 6 months after discontinuation from study medication in case of premature discontinuation. (Note: Hormone-based contraception alone may not be reliable when taking IMP; therefore, hormone-based contraceptives alone cannot be used by female participants to prevent pregnancy).
9. Male participants who are having heterosexual intercourse with females of child-bearing potential are required to use one of the following birth control methods during their participation in the trial and for 12 weeks after their last dose of study medication to prevent pregnancy:

   * a double barrier method which can include a male condom, diaphragm, cervical cap, or female condom; or
   * a barrier method combined with hormone-based contraceptives or an intra-uterine device for the female partner.

The use of the above mentioned birth control method does not apply if the male participant has been vasectomised or has had a bilateral orchidectomy minimally one month prior to screening, or is not heterosexually active, or practice sexual abstinence or if the female sexual partner has had a bilateral oophorectomy and/or hysterectomy or has been postmenopausal for at least 12 consecutive months.

Exclusion Criteria

Medical History

1. Evidence of clinically significant (as judged by the investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
3. A history of previous TB.
4. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
5. History of allergy to the IMP or related substances, including a known allergy to any fluoroquinolone antibiotic, history of tendinopathy associated with quinolones or suspected hypersensitivity to any rifamycin antibiotics.
6. Isoniazid-resistant and Rifampicin-resistant bacteria detected with a sputum specimen collected within the pre-treatment period and tested at the study laboratory.
7. Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the participant.
8. HIV infected participants:

   1. having a CD4+ count <300 cells/µL;
   2. or having received antiretroviral therapy medication within the last 90 days;
   3. or having received oral or intravenous antifungal medication within the last 90 days;
   4. or with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB).
9. Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
10. Significant cardiac arrhythmia requiring medication.
11. Participants with the following at screening:

    1. Marked prolongation of QT/QTc interval, e.g., confirmed demonstration of QTcF (Fridericia correction) or QTcB (Bazett correction) interval >450 ms at screening;
    2. History of additional risk factors for Torsade de Pointes, e.g., heart failure, hypokalemia, family history of Long QT Syndrome;
    3. Use of concomitant medications that prolong the QT/QTc interval (see exclusion criterion 22 as well as list of disallowed medication in Section 4.7.2);
    4. Pathological Q waves (defined as >40ms or depth >0.4-0.5mV);
    5. ECG evidence of ventricular pre-excitation;
    6. ECG evidence of complete or incomplete left bundle branch block or right bundle branch block;
    7. ECG evidence of second or third degree heart block;
    8. Intraventricular conduction delay with QRS duration >120ms;
    9. Bradycardia as defined by sinus rate <50bpm.
12. Females who are pregnant, breast-feeding, or planning to conceive a child within 6 months of cessation of treatment.
13. Males planning to conceive a child within twelve weeks of cessation of treatment.
14. History and/or presence (or evidence) of neuropathy or epilepsy.
15. Diabetes Mellitus requiring insulin.
16. History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination.
17. For males, any evidence or history of a clinically significant abnormality in the reproductive system, including but not limited to the following: serum testosterone, luteinizing hormone (LH), and/or follicle-stimulating hormone (FSH) levels outside the laboratory reference range. An evaluation resulting in an isolated abnormal value (i.e., only 1 of the 3 hormones is abnormal) may be repeated using a morning (ideally, 8am) serum specimen. If the laboratory value on the repeat specimen is outside the laboratory reference range, unless the result is deemed not clinically significant by the Investigator in consultation with the Sponsor Medical Monitor, the participant should be excluded.

    Specific Treatments
18. Previously received treatment with TMC207 or PA-824 as part of a clinical trial.
19. Treatment received with any drug active against MTB within the 3 months prior to Visit 1 (e.g. isoniazid, ethambutol, amikacin, cycloserine, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, fluoroquinolones, thioamides, metronidazole).
20. Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.
21. Any disease or conditions in which any of the medicinal products listed in the section pertaining to prohibited medications is used.
22. Concomitant use of any drug known to prolong QTc interval (including amiodarone, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine). The exception is moxifloxacin which is one of the drugs being evaluated in this study, with extensive ECG monitoring to help ensure patient safety.
23. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (such as quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan). Exceptions may be made for participants that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period before administration of IMP equivalent to at least 5 half-lives of that drug or substance.
24. Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine) within 30 days prior to dosing.
25. Use of systemic glucocorticoids within one year prior to dosing.

    Based on Laboratory Abnormalities
26. Participants with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):

    1. creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    2. lipase grade 3 or greater (>2.0 x ULN);
    3. hemoglobin grade 4 (<6.5 g/dL);
    4. platelets grade 2 or greater (under 50x109 cells/L);
    5. serum potassium grade 2 or greater (<3.5 mEq/L);
    6. aspartate aminotransferase (AST) grade 3 (≥3.0 x ULN) to be excluded;
    7. alanine aminotransferase (ALT) grade 3 (≥3.0 x ULN) to be excluded;
    8. alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 x ULN) must be discussed with the sponsor Medical Monitor;
    9. total bilirubin grade 3 or greater (>2.0 x ULN, or >1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (>1.50 x ULN, or >1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with the sponsor Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diacon, Principal Investigator — Karl Bremer Hospital, Cape Town South africa
Locations (2):
- South Africa (2):
  - Centre for Tuberculosis Research Innovation, UCT Lung Institute, Cape Town
  - Task Applied Science, Karl Bremer Hospital, Cape Town

REFERENCES:
- [Result] Diacon AH, Dawson R, von Groote-Bidlingmaier F, Symons G, Venter A, Donald PR, van Niekerk C, Everitt D, Winter H, Becker P, Mendel CM, Spigelman MK. 14-day bactericidal activity of PA-824, bedaquiline, pyrazinamide, and moxifloxacin combinations: a randomised trial. Lancet. 2012 Sep 15;380(9846):986-93. doi: 10.1016/S0140-6736(12)61080-0. Epub 2012 Jul 23. PMID 22828481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from outpatient clinics and were admitted to the hospital for the duration of the study at one of 2 centers in Capetown, South Africa. The study was conducted between October 2010 and August 2011. Patients aged 18 and 65 years with newly diagnosed smear-positive pulmonary TB were recruited and randomized centrally.
Pre-assignment Details: In the screening period, TB treatment was not provided while baseline sputum was collected/tested. This period was up to 9 days, up to 6 days screening followed by 3 days baseline sputum collection. Hospitalization during this time was left to investigator discretion. 173 patients were screened and 88 patients discontinued before randomization.
Groups:
- TMC207: TMC207 administered once daily as 100mg tablets for a total daily dose of 700mg on Day 1; 500mg on Day 2; 400mg on Days 3-14 plus pyrazinamide placebo tablets (matched to pyrazinamide tablets) administered once daily on Days 1-14 dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day
- TMC207 and Pyrazinamide: TMC207 administered once daily as 100mg tablet for total daily dose of 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus pyrazinamide administered once daily on Days 1-14 as 500mg tablets dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day
- PA-824 and Pyrazinamide: PA-824 administered once daily as 200mg tablets for a total daily dose of 200mg on Days 1-14, pyrazinamide administered once daily on Days 1-14 as 500mg tablets dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day, and moxifloxacin placebo tablets (matched to moxifloxacin tablets) administered once daily on Days 1-14
- PA-824 and Moxifloxacin and Pyrazinamide: PA-824 administered once daily as 200mg tablets for a total daily dose of 200mg on Days 1-14, pyrazinamide administered once daily on Days 1-14 as 500mg tablets dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day, and moxifloxacin administered once daily as 400mg tablets for a total daily dose of 400mg on Days 1-14
- Rifafour e-275 mg: Rifafour e-275 administered once daily on Days 1-14 with each tablet containing 150mg rifampicin, 75mg isoniazid, 400mg pyrazinamide, and 275mg ethambutol and dosed by weight as follows: 30kg - 37kg received 2 tablets/day; 38kg - 54kg received 3 tablets/day; 55kg - 70kg received 4 tablets/day; > or = 71kg received 5 tablets/day
- TMC207 and PA-824: TMC207 administered once daily as 100mg tablet for total daily dose of 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus PA-824 administered once daily as 200mg tablets for a total daily dose of 200mg on Days 1-14
Period: Treatment Period
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Started | 15 | 15 | 15 | 15 | 10 | 15
Completed | 14 | 14 | 14 | 12 | 10 | 14
Not Completed | 1 | 1 | 1 | 3 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 3 | 0 | 1
Period: Follow up Period
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Started | 14 | 14 | 14 | 12 | 10 | 14
Completed | 14 | 14 | 14 | 12 | 10 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PA-824 and Moxifloxacin and Pyrazinamide: PA-824 administered once daily as 200mg tablets and pyrazinamide administered once daily in 500mg tablets dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day and moxifloxacin administered once daily as 400mg tablets for a total daily dose of 400mg on Days 1-14
- Rifafour e-275 mg: Rifafour e-275 administered once daily with each tablet containing 150mg rifampicin, 75mg isoniazid, 400mg pyrazinamide, and 275mg ethambutol and dosed by weight as follows: 30kg - 37kg received 2 tablets/day; 38kg - 54kg received 3 tablets/day; 55kg - 70kg received 4 tablets/day; > or = 71kg received 5 tablets/day
- Total: Total of all reporting groups
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 15 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 10 | 15 | 85
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (11.60) | 29.1 (8.67) | 29.7 (8.93) | 28.3 (9.34) | 27.0 (6.63) | 33.3 (8.47) | 30.0 (9.13)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 4 | 4 | 22
  Male | 11 | 12 | 11 | 12 | 6 | 11 | 63
Region of Enrollment [Number; unit: participants]
  South Africa | 15 | 15 | 15 | 15 | 10 | 15 | 85

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-14).
Description: Log10 CFU rates of change were calculated for each individual patient from the slopes β1 and β2 of the bi-linear regression fitted to the data for each individual patient (log10CFU versus Day). Mean log10 CFU changes from baseline were compared. A higher slope value indicates a greater change in log10 CFU from baseline. Note that to facilitate interpretation the sign of these slopes are reversed for logCFU. A positive slope value therefore indicates a reduction in log10 CFU from baseline.
Time Frame: 14 consecutive days of treatment
Population: In the case of patient dropout, their patient data were included in the analyses as long as enough points were recorded to allow curve fitting. The number of patients analyzed for this outcome was 80.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Number analyzed (Participants) | 14 | 15 | 14 | 13 | 10 | 14
log10CFU/ml/day | 0.061 (0.068) | 0.131 (0.102) | 0.154 (0.040) | 0.233 (0.128) | 0.140 (0.094) | 0.114 (0.050)

2. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-2).
Description: as for outcome 1
Time Frame: Day 0-2
Population: In the case of patient dropout, their patient data were included in the analyses as long as enough points were recorded to allow curve fitting. The number patients analyzed for this measure was 84.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 14
log10CFU/ml/day | -0.022 (0.121) | 0.079 (0.167) | 0.170 (0.082) | 0.315 (0.133) | 0.177 (0.188) | 0.114 (0.149)

3. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 2-14).
Description: as for outcome 1
Time Frame: Day 2-14
Population: In the case of patient dropout, their patient data were included in the analyses as long as enough points were recorded to allow curve fitting. The number of patients analyzed for this measure was 80.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Groups:
- TMC207 and Pyrazinamide: MC207 administered once daily as 100mg tablet for total daily dose of 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus pyrazinamide administered once daily on Days 1-14 as 500mg tablets dosed by weight as follows: < or = 55kg 2 tablets/day; >55kg to 75kg 3 tablets/day; >75kg 4 tablets/day
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Number analyzed (Participants) | 14 | 15 | 14 | 13 | 10 | 14
log10CFU/ml/day | 0.076 (0.069) | 0.143 (0.109) | 0.148 (0.043) | 0.222 (0.130) | 0.135 (0.103) | 0.114 (0.047)

4. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Change of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 7-14).
Description: as for outcome 1
Time Frame: Day 7-14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Number analyzed (Participants) | 14 | 15 | 14 | 13 | 10 | 14
log10CFU/ml/day | 0.123 (0.097) | 0.152 (0.120) | 0.124 (0.080) | 0.175 (0.146) | 0.136 (0.102) | 0.114 (0.069)

5. Secondary Outcome: Rate of Change in Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 0-14)
Description: The TTP was measured in the Mycobacterial Growth Indicator Tube (MGIT) (Bactec MGIT960) automated liquid culture system from overnight sputum. TTP rates of change were calculated for each individual patient from the slopes β1 and β2 of the bi-linear regression fitted to the data for each individual patient (TTP versus Day).
Time Frame: 14 Days
Population: In the case of patient dropout, their patient data were included in the analyses as long as enough points were recorded to allow curve fitting. The number of patients analyzed for this measure was 81.
Measure: Mean (Standard Deviation); unit: time (h) to positive per day
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Number analyzed (Participants) | 14 | 15 | 14 | 13 | 10 | 15
time (h) to positive per day | 5.414 (3.523) | 9.970 (6.987) | 8.805 (3.468) | 18.482 (22.582) | 11.841 (3.932) | 5.855 (2.785)

ADVERSE EVENTS:
Groups:
- TMC207: TMC207 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus pyrazinamide placebo
- TMC207 and Pyrazinamide: TMC207 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus pyrazinamide (dosed by weight)
- PA-824 and Pyrazinamide: PA-824 200mg and pyrazinamide (dosed by weight)and moxifloxacin placebo
- PA-824 and Moxifloxacin and Pyrazinamide: PA-824 200 mg and pyrazinamide (dosed by weight) and moxifloxacin 400 mg
- Rifafour e-275 mg: Rifafour e-275 275 mg
- TMC207 and PA-824: TMC207 700 mg Day 1; 500mg Day 2; 400mg Days 3-14 plus PA-824 200 mg
Arm/Group | TMC207 | TMC207 and Pyrazinamide | PA-824 and Pyrazinamide | PA-824 and Moxifloxacin and Pyrazinamide | Rifafour e-275 mg | TMC207 and PA-824
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 1/15 | 0/10 | 1/15
Other Adverse Events (participants affected / at risk) | 7/15 | 6/15 | 7/15 | 8/15 | 5/10 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMC207 (N=15) | TMC207 and Pyrazinamide (N=15) | PA-824 and Pyrazinamide (N=15) | PA-824 and Moxifloxacin and Pyrazinamide (N=15) | Rifafour e-275 mg (N=10) | TMC207 and PA-824 (N=15)
Worsening of Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurocysticercosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMC207 (N=15) | TMC207 and Pyrazinamide (N=15) | PA-824 and Pyrazinamide (N=15) | PA-824 and Moxifloxacin and Pyrazinamide (N=15) | Rifafour e-275 mg (N=10) | TMC207 and PA-824 (N=15)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type I diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
With the small sample, individual results can influence overall results. Comparison between groups and studies is difficult. The ability to assign AEs to a particular compound is limited. The value of EBA studies for predicting relapse is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information given to the Investigator by the Sponsor shall not be published/disclosed to a third party, other than to IEC/IRB, within the understanding of the confidentiality, without the prior written consent of the Sponsor. Results of this research will be submitted for publication as soon as feasible upon completion of the study in the form of a joint publication(s) between the Sponsor and Investigator(s), including site clinical and laboratory investigators, as appropriate.